CLINICAL TRIAL: NCT06112457
Title: Anxiety and Depression Among Gendarmes Posted to French Guiana (TAD-GENDGF)
Brief Title: Anxiety and Depression Among Gendarmes Posted to French Guiana
Acronym: TAD-GENDGF
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Direction Centrale du Service de Santé des Armées (Other)
Responsible Party: Sponsor
Other Study IDs: 2022PPRC07; 2023-100889-36 (Other: IDRCB)
Record Dates: First submitted 2023-10-26; First posted 2023-11-01 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Anxiety Depression Disorder
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Survey — Anonymous self-administered questionnaire

SUMMARY:
This is a mixed-method, single-center study involving two concurrent phases: a quantitative phase with an anonymous self-administered questionnaires, and a qualitative phase with individual contextual interviews and a focus group. The hypothesis underlying this study is that isolated postings are a risk factor for anxiety-depressive disorders. The aim of this study is to provide new information to help propose targeted prevention and health promotion measures.

ELIGIBILITY:
Inclusion Criteria:

* Gendarme in active position
* Age over 18
* Assignment in French Guiana for more than 6 months at the time of the study
* Not opting for study participation

Exclusion Criteria:

* Previously diagnosed psychiatric condition
* People with a reading/writing disability in the French language
* Major incapacity

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healthy volunteer
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2023-11 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Prevalence of anxiety-depressive disorders according to posting site. | Through study completion (6 months)
  Comparison of the prevalence of anxiety-depressive disorders among gendarmes posted to French Guiana according to their posting site.

SECONDARY OUTCOMES:
Factors associated with the presence of an anxiety-depressive disorder | Through study completion (6 months)
  Evaluate factors associated with the presence of an anxiety-depressive disorder, both overall and by type of disorder

CONTACTS AND LOCATIONS:
Locations (1):
- DIASS Guyane, Cayenne, Guyane, French Guiana

IPD SHARING:
Plan to Share IPD: Undecided